CLINICAL TRIAL: NCT03408015
Title: Effects of Xiidra on Closed Eye Tear Film Leukocytes in Dry Eye Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study timing was poor.
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Kelly Nichols, Dean, Principal Investigator, UAB School of Optometry, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 300001139
Record Dates: First submitted 2018-01-17; First posted 2018-01-23 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Ocular Discomfort; Ocular Inflammation; Dry Eye; Contact Lens Complication; Keratoconjunctivitis Sicca
Keywords: dry eye disease; neutrophil; T cell; lifitegrast; contact lens discomfort; ocular surface homeostasis
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — lifitegrast

STUDY DESIGN:
Intervention Model Description: Three groups of individuals will be recruited: asymptomatic non-contact lens wearers; symptomatic non-contact lens wearers, with dry eye disease; symptomatic contact lens wearers, with contact lens discomfort. All three groups will receive the same Xiidra treatment for the complete study duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal, asymptomatic non-lens wearers (Experimental): Lifitegrast ophthalmic solution, 5.0%. Dosage: 1 drop in each eye, twice daily: once in the morning and once before bed.
  Interventions: Drug: Lifitegrast
- Dry eye subjects, non-lens wearers (Experimental): Lifitegrast ophthalmic solution, 5.0%. Dosage: 1 drop in each eye, twice daily: once in the morning and once before bed.
  Interventions: Drug: Lifitegrast
- Contact lens wearers with discomfort (Experimental): Lifitegrast ophthalmic solution, 5.0%. Dosage: 1 drop in each eye, twice daily: once in the morning and once before bed.
  Interventions: Drug: Lifitegrast

INTERVENTIONS:
Drug: Lifitegrast — Lifitegrast ophthalmic solution, 5.0%. 1 drop instilled into each eye once in the morning and once before bed.
  Other Names: Xiidra

SUMMARY:
Every night during sleep, there is an accumulation of white blood cells in the closed eye. The closed eye white blood cells are predominantly neutrophils, but there is a small population (3%) of T cells. The effects of these closed eye white blood cells on dry eye disease pathogenesis have yet to be fully elucidated, but preliminary evidence suggests that closed eye neutrophils may have an associated hyperactivity and increased degranulation in dry eye disease that could contribute to epithelial instability. As an anti-T cell therapy, Xiidra offers an opportunity to better understand how the closed eye white blood cells are recruited and activated. This study also seeks to verify the proposed mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an informed consent and HIPAA privacy document
* Greater than 18 years of age at time of informed consent
* Able and willing to follow protocol instructions
* Capable of performing at-home eye wash
* Must be willing to drop off samples and comply with study visit procedures
* For contact lens wearers, must wear lenses at least four hours per day, four days per week

Exclusion Criteria:

* Current cigarette smokers
* Current participation in any investigational drug or device study. If subjects choose to participate in another investigational drug or device study, they will be discontinued from this study protocol.
* Current pregnancy or nursing as indicated by self-report. While not a safety issue, pregnancy or nursing influences the biochemical composition of the tear film.
* Any systemic health conditions that alter tear film physiology
* A history of ocular surgery within the past 12 months
* Any active ocular infection or inflammation
* Any present use of Accutane or ocular medications
* Any history of significant adverse reaction to lifitegrast or other components of the drug product, or contraindication to the use of lifitegrast or other components of the drug product
* Any prior exposure to lifitegrast.
* For normal and dry eye subjects, any history of contact lens wear within the past three months.
* For contact lens wearers, any change of soft contact lens brand or care solutions within 30 days prior to screening or any anticipation of changing current type/brand of contact lenses or care solutions throughout the 84 day study
* Any condition, which in the examiner's opinion, may put the subject at significant risk, confound study results, or interfere with their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the total number of T cells recovered from the closed eye to day 84 | Baseline to day 84
  Subjects will be trained and required to collect their closed eye tears at home, using a gentle saline rinse of the ocular surface. Enumeration of recovered T cells will be performed by flow cytometry.

SECONDARY OUTCOMES:
Change from baseline in the total number of neutrophils recovered from the closed eye to day 84. | Baseline to day 84.
  Subjects will be trained and required to collect their closed eye tears at home, using a gentle saline rinse of the ocular surface. Enumeration of recovered neutrophils will be performed by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly K Nichols, OD MPH PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No